CLINICAL TRIAL: NCT06486077
Title: Full Title: Metabolic Health 1: Power Line Evaluation; Effect Size Determination
Brief Title: Metabolic Health 1: Power Line Evaluation; Effect Size Determination
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nature's Sunshine Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NSP-CT-021
Record Dates: First submitted 2024-06-18; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Metabolic Health

STUDY DESIGN:
Intervention Model Description: Open Label, Single Arm Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Power Line Program (Experimental): Daily supplementation with Power Line program consisting of 4 nutritional supplements: a meal replacement shake, a vegetable based green drink, a vascular health product, and a pre-meal fiber supplement. Subjects will maintain their current lifestyle (specifically diet, exercise, and nutritional supplements) during intervention.
  Interventions: Dietary Supplement: Power Line Program

INTERVENTIONS:
Dietary Supplement: Power Line Program — Power Line program consisting of 4 nutritional supplements: a meal replacement shake, a vegetable based green drink, a vascular health product, and a pre-meal fiber supplement

SUMMARY:
The primary goal of this study is to demonstrate the safety and tolerability of the Power Line program, an integrated, whole-food supplement system. Secondarily, it is desired to determine the effect size of this program on maintenance of markers of metabolic health, with a particular emphasis on insulin sensitivity and dyslipidemia.

DETAILED DESCRIPTION:
From 1960-1962, 13.4% of adults (aged 20-74) in the United States were considered obese (BMI 30.0-39.9) and less than 1% of adults were considered severely obese (BMI 40.0 and above). By 2018 the number of obese adults had risen to 42.8% and severely obese adults had risen to 9.6% of the population . By 2030 it is estimated that 48.9% of adults will be considered obese and 24.2% of adults will be considered severely obese, with severe obesity becoming the most common BMI category for women, low-income adults, and non-Hispanic black adults . Metabolic syndrome, diabetes, heart disease, and other non-communicable diseases are on the rise, particularly among children, women, and the lower socioeconomic classes . There is a strong correlation between diet, particularly the increased consumption of highly processed foods and underconsumption of vegetables and poorer metabolic health outcomes . While physical activity is known to be a major component of metabolic health , improving one's diet, even in the absence of increased physical activity, can have an important impact on improving metabolic health .

Metabolic health, for the purpose of this study, will be defined in terms of the 5 cardiovascular risk factors associated with metabolic syndrome. The risk factors associated with metabolic syndrome are elevated fasting blood glucose level, obesity (as measured by waist circumference), elevated triglycerides, elevated blood pressure, and low HDL cholesterol . There is a process by which long-term lifestyle choices lead to reduced metabolic health, then metabolic syndrome, then other lifestyle diseases such as type II diabetes. Poor food choices and lack of physical activity give rise to chronically elevated insulin levels, a slow increase in insulin resistance, and eventual insulin insensitivity and even the complete inability to produce insulin . Throughout much of this decline in metabolic health, the process is reversible by improving lifestyle choices .

While there is significant literature that demonstrates the impact of diet on metabolic health, the literature tends to focus on interventions that involve a change to a specific type of diet (i.e. the Mediterranean diet or keto diet), changes in specific macronutrient consumption (i.e. increased protein consumption leading to improved body composition), or the introduction of specific phytonutrients or botanical ingredients . Moreover, studies on dietary interventions for metabolic health, particularly those that involve supplementation, are often confounded with factors such as additional changes in diet or exercise level . Based on the current literature, it is possible to understand how specific macronutrients and micronutrients can potentially interact to support metabolic health, but controlled study on a complete supplement system that utilizes the current literature as a foundation for its genesis is lacking.

ELIGIBILITY:
Inclusion Criteria:

Generally healthy Female, Male and Non-Binary adults, 18-64 years of age (Inclusive)

Body Mass Index (BMI): 28.0-34.9 kilograms/meters2 (kg/m2) (Inclusive)

Preference given to individuals having a minimum of two of the following markers of metabolic imbalance: fasting blood glucose ≥ 100 milligrams/deciliter (mg/dl), serum triglycerides (TG) >100 mg/dl, serum high density lipoprotein - cholesterol (HDLc) (male sex < 40 mg/dl, female sex < 50 mg/dl), elevated blood pressure (systolic ≥ 120 and /or diastolic ≥ 80), elevated waist circumference (male sex ≥ 40 inches, female sex ≥ 35 inches)

Willing to maintain a consistent diet (including medications, vitamins, and supplements) and lifestyle routine throughout the study.

Willing to give written informed consent to participate in the Study.

Exclusion Criteria:

A serious, unstable illness including cardiac, hepatic, renal, gastrointestinal, respiratory, endocrinologic, neurologic, immunologic/rheumatological, or oncological/hematologic disease.

Allergies related to ingredients in study products

Known infection with HIV, TB or Hepatitis B or C.

POCBP: Not using effective contraception.

Blood Pressure medications or supplements

Diabetes medications or supplements

Cholesterol/Triglyceride lowering medications or supplements

Currently taking nutritional supplements judged by the study coordinator to negate or camouflage the effects of the study products

Use of Narcotics during the last 30 days

Use of Anticoagulants during last 30 days

Use of Corticosteroids during the last 30 days

Use of controlled substances on a recreational basis during the last 30 days.

Consumption of more than 3 alcoholic beverages per day. One beverage is a 5-ounce glass of wine, 12 ounces of beer, or one ounce of hard liquor.

Inability to comply with Study and/or follow-up visits.

Any concurrent condition (including clinically significant abnormalities in medical history, physical examination, or laboratory evaluations) which, in the opinion of the PI, would preclude safe participation in this study or interfere with compliance.

Any sound medical, psychiatric, and/or social reason which, in the opinion of the PI, would preclude safe participation in this Study or interfere with compliance.

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with supplementation-related adverse events (AEs) as assessed by Common Terminology Criteria for Adverse Events v4.0 (CTCAE v4.0). | 90 days
  Data collection at individual study visits (visit 1- baseline, visit 2 - Day 30, visit 3 - Day 60 and visit 4 - Day 90) will be used to assess participants for supplementation program-related adverse events. Subjects with ongoing AEs may be followed until resolution at the discretion of the PI.

SECONDARY OUTCOMES:
Number of participants with treatment-related changes in basic safety labs | 90 days
  Phlebotomy will be conducted at individual visits (visit 1- baseline, visit 3 - Day 60 and visit 4 - Day 90). Comprehensive Metabolic Panels and Complete Blood Counts will be assessed for treatment-related change from baseline
Number of participants with treatment-related changes in vital signs | 90 days
  Blood pressure, respiratory rate and pulse rate will be monitored at individual visits (visit 1- baseline, visit 2 - Day 30, visit 3 - Day 60 and visit 4 - Day 90). Collected data will be assessed for treatment-related change from baseline
Change in anthropometric measures compared to baseline | 90 days
  Body composition analyses ( Muscle-fat, obesity, segmental lean, ECW/TBW), height, hip circumference, waist circumference, weight and BMI will be monitored at individual visits (visit 1- baseline, visit 2 - Day 30, visit 3 - Day 60 and visit 4 - Day 90). Collected data will be assessed for treatment-related change from baseline.
Change in urinalysis measures compared to baseline | 90 days
  Uninalysis will be conducted using Medline Urinalysis Reagent Strips at individual visits (visit 1 -baseline, visit 3 - Day 60 and visit 4 - Day 90). Collected data will be assessed for treatment-related change from baseline.
Change in Hemoglobin A1c in percentage compared to baseline | 90 days
  Hemoglobin A1c in percentage will be measured at individual visits (visit 1- baseline, visit 3 - Day 60 and visit 4 - Day 90). Collected data will be assessed for treatment-related change from baseline.
Change in fasting Insulin compared to baseline | 90 days
  Fasting Insulin will be measured at individual visits (visit 1- baseline, visit 3 - Day 60 and visit 4 - Day 90). Collected data will be assessed for treatment-related change from baseline.
Change in Triglycerides compared to baseline | 90 days
  Triglycerides will be measured at individual visits (visit 1- baseline, visit 3 - Day 60 and visit 4 - Day 90). Collected data will be assessed for treatment-related change from baseline.
Change in Total Cholesterol compared to baseline | 90 days
  Total Cholesterol will be measured at individual visits (visit 1- baseline, visit 3 - Day 60 and visit 4 - Day 90). Collected data will be assessed for treatment-related change from baseline.
Change in LDL-Cholesterol compared to baseline | 90 days
  LDL-Cholesterol will be measured at individual visits (visit 1- baseline, visit 3 - Day 60 and visit 4 - Day 90). Collected data will be assessed for treatment-related change from baseline
Change in oxidized LDL-Cholesterol compared to baseline | 90 days
  Oxidized LDL-Cholesterol will be measured at individual visits (visit 1- baseline, visit 3 - Day 60 and visit 4 - Day 90). Collected data will be assessed for treatment-related change from baseline.
Change in HDL-Cholesterol compared to baseline | 90 days
  HDL-Cholesterol will be measured at individual visits (visit 1- baseline, visit 3 - Day 60 and visit 4 - Day 90). Collected data will be assessed for treatment-related change from baseline.
Changes in self-perceived health using a Health questionaire | 90 days
  The study staff will review the Health questionnaire at individual visits (visit 1- baseline, visit 2 - Day 30, visit 3 - Day 60 and visit 4 - Day 90).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Lamb, MD, Principal Investigator — Natures Sunshine
Locations (1):
- The Hughes Center for Research and Innovation, Lehi, Utah, United States

IPD SHARING:
Plan to Share IPD: No